CLINICAL TRIAL: NCT06498882
Title: Impact of Press Needle Acupoint Stimulation Combined With Breast Massage on the Initiation of Lactogenesis II: A Randomized Controlled Trial
Brief Title: Press Needle Acupoint Stimulation Combined With Breast Massage on the Initiation of Lactogenesis II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qingdao Municipal Hospital (Other)
Responsible Party: Principal Investigator, Jia Qiao, RN, Qingdao Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Grant No.(2023LinShenZi No.122
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Lactation Induced
Keywords: press needle; acupoint stimulation; breast massage; lactogenesis II; breastfeeding sessions; breast milk composition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- press needle acupoint stimulation combined with breast massage group (Experimental): On the basis of the routine care, press needle acupoint stimulation and breast massage were administered to the intervention group
  Interventions: Other: Press Needle Acupoint Stimulation Combined with Breast Massage; Other: routine care
- control group (Other): Control group received routine care
  Interventions: Other: routine care

INTERVENTIONS:
Other: Press Needle Acupoint Stimulation Combined with Breast Massage — Press needle acupoint stimulation and breast massage were administered. Key press needle acupoints were identified for selection: Dan zhong (RN17), bilateral Ru gen (ST18), bilateral Shao ze (SI1), bilateral Zu san li (ST36) and bilateral San yin jiao (SP6). The areas were sterilized with 75% alcohol before installing 0.22*1.55mm press needles. Within 4-6 hours post-surgery, mothers received acupoint stimulation through needle pressing. This procedure was administered by nurses who had undergone six-month standardized training in traditional Chinese medicine techniques. Instructions were then given to mothers and their family members to stimulate the acupoints pulsatively every 3-4 hours for 20-30 minutes per session, removing the press needles after 24 hours. Additionally, a specialized nurse massaged the back, both breast areas, and armpits for 10-15 minutes, three times daily over three days, using a circular and oscillating breast massage device.
  Arms: press needle acupoint stimulation combined with breast massage group
Other: routine care — Very early skin-to-skin contact was initiated by researchers within 30 to 40 minutes after birth, with newborns, optionally wearing caps, being placed on the mothers' chests. Mothers were encouraged to breastfeed 8 to 10 times per day to ensure steady milk production. It was ensured by researchers that mothers completely emptied one breast before switching to the other to maintain cleanliness. Additionally, mothers were guided by researchers on maintaining a well-balanced diet, achieving emotional stability, and securing adequate sleep to facilitate effective breastfeeding.

SUMMARY:
This RCT aimed to rigorously evaluate the combined effects of press needle acupuncture and breast massage on accelerating the onset of lactogenesis II, thereby optimizing breastfeeding outcomes and maternal health post-cesarean delivery. It involved 136 mothers who had cesarean sections at this facility along with their healthy single-born infants.

Control group received routine care. On the basis of the control group, press needle acupoint stimulation and breast massage were administered to the intervention group. The main outcome indicators included the sensation of milk coming in, defined as the time to stage II lactogenesis. Additionally, milk quality was assessed 72 hours after birth, focusing on the content of protein, fat, lactose, minerals, and water. Secondary outcomes tracked include the number of breastfeeding sessions within the first 72 hours, the milliliters of formula provided to the infant during this period, and the percentage of mothers exclusively breastfeeding after 72 hours.

DETAILED DESCRIPTION:
This RCT aimed to rigorously evaluate the combined effects of press needle acupuncture and breast massage on accelerating the onset of lactogenesis II, thereby optimizing breastfeeding outcomes and maternal health post-cesarean delivery. It involved 136 mothers who had cesarean sections at this facility along with their healthy single-born infants.

Control group: Very early skin-to-skin contact was initiated by researchers within 30 to 40 minutes after birth, with newborns, optionally wearing caps, being placed on the mothers'chests. Mothers were encouraged to breastfeed 8 to 10 times per day to ensure steady milk production. Additionally, mothers were guided by researchers on maintaining a well-balanced diet, achieving emotional stability, and securing adequate sleep to facilitate effective breastfeeding.

Intervention group: On the basis of the control group, press needle acupoint stimulation and breast massage were administered to the intervention group.

Primary Outcome Measurement: The main outcome indicators included the sensation of milk coming in, defined as the time to stage II lactogenesis. Participants were asked to report the approximate time they noticed their breasts feeling "noticeably fuller" using a numeric scale: 1 indicated "no change since giving birth", 3 denoted "noticeably fuller", and 5 represented "uncomfortably full" (Lian et al., 2022). Additionally, milk quality was assessed 72 hours after birth, focusing on the content of protein, fat, lactose, minerals, and water.

Secondary Outcome Measurements: Secondary outcomes tracked include the number of breastfeeding sessions within the first 72 hours (breastfeeds, first 24 h, 24-48 h, 48-72 h), the milliliters of formula provided to the infant during this period (formula fed to infant, first 24 h, 24-48 h, 48-72 h), and the percentage of mothers exclusively breastfeeding after 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Mothers ≥18 years old
* Expecting their first live-born child via cesarean delivery
* Having a singleton pregnancy
* Intending to breastfeed with no major contraindications like hepatitis B, HIV, or other infectious diseases
* Having newborns with Apgar scores above 8 at 1 and 5 minutes, robust sucking reflex, and no neonatal transfer required
* Able to understand and respond to questions
* Accessible for follow-up via telephone or WeChat

Exclusion Criteria:

* Mothers having previous breast surgeries like biopsies or augmentations
* Having nipple inversions that complicate breastfeeding; (c) taking medications affecting lactation
* Experiencing severe perinatal complications, such as serious pre-eclampsia or grade 3 or higher cardiac issues per NYHA standards
* Having severe local skin damage at the acupoint and massage sites
* Having newborns with critical conditions like cardiopulmonary insufficiency, galactosemia, or phenylketonuria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
time to stage II lactogenesis | 0-96 hours after delivery
  The main outcome indicators included the sensation of milk coming in, defined as the time to stage II lactogenesis. Participants were asked to report the approximate time they noticed their breasts feeling 'noticeably fuller' using a numeric scale: 1 indicated 'no change since giving birth, '3 denoted 'noticeably fuller,' and 5 represented 'uncomfortably full' (Lian et al., 2022).
milk quality | 72 hours after delivery
  Milk quality was assessed 72 hours after birth, focusing on the content of protein, fat, lactose, minerals, and water.

SECONDARY OUTCOMES:
number of breastfeeding sessions | a) 0-24 hours, 24-48 hours, 48-72 hours after delivery
  Secondary outcomes tracked include the number of breastfeeding sessions within the first 72 hours (breastfeeds, 0-24 hours, 24-48 hours, 48-72 hours)
milliliters of formula provided to the infant | 0-24 hours, 24-48 hours, 48-72 hours after delivery
  Secondary outcomes tracked include the milliliters of formula provided to the infant during this period (formula fed to infant, 0-24 hours, 24-48 hours, 48-72 hours)
percentage of mothers exclusively breastfeeding | 72 hours after delivery
  Secondary outcomes tracked include the percentage of mothers exclusively breastfeeding after 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Shan Huan, Bachelor, Study Director — Qingdao Municipal Hospital; Jia Qiao, Master, Principal Investigator — Qingdao Municipal Hospital
Locations (1):
- Qingdao Municipal Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Sharing study protocol.
Supporting Information: Study Protocol
Time Frame: 31/08/2025 to 31/08/2018
Access Criteria: On reasonable request

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Background] Becker GE, Smith HA, Cooney F. Methods of milk expression for lactating women. Cochrane Database Syst Rev. 2016 Sep 29;9(9):CD006170. doi: 10.1002/14651858.CD006170.pub5. PMID 27684560
- See also: view only — https://www.kdocs.cn/l/ct2MPLDPYLoR
- Available data/document: Individual Participant Data Set — https://kdocs.cn/l/cftB6eP0xNOu — The authors have full control of all primary data and that they agree to allow other researchers to review their data if requested.